CLINICAL TRIAL: NCT07047612
Title: A Phase II/III Randomized, Double-blind, Placebo-controlled, Parallel Group, Adaptive Design, Multi-center Study to Evaluate the Efficacy and Safety of ICP-332 in Subjects With Non-segmental Vitiligo
Brief Title: ICP-332 in Subjects With Non-segmental Vitiligo
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICP-CL-00607
Record Dates: First submitted 2025-06-23; First posted 2025-07-02 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-04

CONDITIONS: Non Segmental Vitiligo

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- ICP-332 dose A（Phase2） (Experimental)
  Interventions: Drug: ICP-332 Tablets
- Placebo（Phase2） (Placebo Comparator)
  Interventions: Drug: ICP-332 Placebo Tablets
- ICP-332 dose B（Phase2:） (Experimental)
  Interventions: Drug: ICP-332 Tablets
- ICP-332 dose A or dose B（Phase3） (Experimental)
  Interventions: Drug: ICP-332 Tablets
- Placebo（Phase3） (Placebo Comparator)
  Interventions: Drug: ICP-332 Placebo Tablets

INTERVENTIONS:
Drug: ICP-332 Tablets — ICP-332 will be administered as tablet
  Arms: ICP-332 dose A or dose B（Phase3）; ICP-332 dose A（Phase2）; ICP-332 dose B（Phase2:）
Drug: ICP-332 Placebo Tablets — ICP-332 Placebo will be administered as tablet
  Arms: Placebo（Phase2）; Placebo（Phase3）

SUMMARY:
This a phase II/III randomized, double-blind, placebo-controlled, parallel group, adaptive design, multi-center study to evaluate the efficacy and safety of ICP-332 in subjects with non-segmental vitiligo。The study consisted an phase 2 part and an phase 3 part.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥18 years and ≤75 years (Phase II portion). Male or female subjects ≥12 years of age and ≤75 years of age, adolescent subjects must weigh ≥40 kg (Phase III portion).
2. Eligible subjects must meet all of the following criteria at screening and baseline:

   1. The clinical diagnosis was non-segmental vitiligo for at least 3 months.
   2. Involvement of BSA≥5%.
   3. Facial involvement BSA≥0.5%.
   4. F-VASI≥0.5 and T-VASI between 5 and 50.
   5. Active or stable non-segmental vitiligo was present at both screening and baseline visits.
3. Women of childbearing potential (WOCBP) and Men must agree to contraception.
4. Before beginning any screening or study specific procedures, subjects must voluntarily sign informed consent.

Exclusion Criteria:

1. Any of the following vitiligo related medical conditions and other skin diseases/conditions.

   a) Subjects had other types of vitiligo (including but not limited to segmental vitiligo and mixed vitiligo) that did not meet the criteria for active or stable vitiligo described in Inclusion criteria 2.
2. History of any clinically major diseases, with the exception of vitiligo.
3. Pregnant or breastfeeding females.
4. The investigator considers that the subject is not suitable for participation in this study for any reason.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 603 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Phase2: Percent change from baseline in facial vitiligo area scoring index (F-VASI) at week 24. | 24 weeks
Phase3: Proportion of subjects achieving F-VASI 75 at Week 52. | 52 weeks

CONTACTS AND LOCATIONS:
Locations (45):
- China (45):
  - The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - The Second Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Chao-yang Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Chongqing Traditional Chinese Medicine Hospital, Chongqing, Chongqing Municipality
  - Union Hospital affiliated to Fujian Medical, Fuzhou, Fujian
  - The First Affiliated Hospital of Fujian Medical, Fuzhou, Fujian
  - Sun Yat-sen Memorial Hospital,Sun Yat-sen University, Guangzhou, Guangdong
  - Deramatology Hospital of Southern Medical Univercity, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Nanyang First People's Hospital, Nanyang, Henan
  - The First Affiliated Hospital of Xinxiang Medical College, Weihui, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Zhengzhou Central Hospital Affiliated to Zhengzhou University, Zhengzhou, Henan
  - Jingzhou Central Hospital, Jingzhou, Hubei
  - Shiyan People's Hospital, Shiyan, Hubei
  - Wuhan NO.1 Hospital(Wuhan Hospital of Traditional Chinese and Western Medicine), Wuhan, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of University Of South China, Hengyang, Hunan
  - The First People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - Hospital for Skin Diseases, Chinese Academy of Medical Sciences, Nanjing, Jiangsu
  - Suzhou Municipal Hospital, Suzhou, Jiangsu
  - Dermatology hospital of jiangxi province, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The first hospital of Jilin Univercity, Changchun, Jilin
  - Shenyang Medical College Affiliated Central Hospital, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong First Medical University Affiliated Dermatology Hospital (Shandong Institute of Dermatology and Venereology, Shandong Dermatology Hospital), Jinan, Shandong
  - Zibo Central Hospital, Zibo, Shandong
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Dermatology Hospital, Shanghai, Shanghai Municipality
  - Shaanxi Provincial People's Hospital, Xian, Shanxi
  - Chengdu Second People's Hospital, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The First Affiliated Hospital Of Kunming Medical University, Kunming, Yunnan
  - Hangzhou Third People's Hospital, Hangzhou, Zhejiang
  - Affiliated Hangzhou First People's Hospital, School of Medicine, Westlake University, Hangzhou, Zhejiang
  - The First Affiliated Hospital Of Ningbo University, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - The Fourth Affiliated Hospital, Zhejiang University School Of Medicine, Yiwu, Zhejiang